CLINICAL TRIAL: NCT00141596
Title: A Study to Investigate the Contribution of Extracellular Fluid Volume Expansion to Drug Resistant Hypertension
Brief Title: Extracellular Fluid in Resistant Hypertension
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient accrual rate
Sponsor: St George's, University of London (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LREC 03.0001
Record Dates: First submitted 2005-08-31; First posted 2005-09-01 (Estimated); Last update posted 2015-06-09 (Estimated); Status verified 2007-05

CONDITIONS: Hypertension
Keywords: Resistant Hypertension; Extracellular Fluid Volume
MeSH Terms: conditions — Hypertension | interventions — Doxazosin; Amiloride; Furosemide

INTERVENTIONS:
Drug: Cardura XL 4 mg bd
Drug: Amiloride 5 mg bd
Drug: Furosemide 40 mg bd

SUMMARY:
The optimal treatment of drug resistant (defined as BP> 140/85 despite three anti-hypertensive drugs including a diuretic) is not well defined. This study aims to test the hypothesis that resistant hypertension is caused by excessive expansion of extracellular fluid volume. A secondary objective is to study which of three different antihypertensive drugs would be most useful in drug resistant hypertension.

DETAILED DESCRIPTION:
Following recruitment subjects will have ECV measured by 51Cr-EDTA determination of GFR, with Brochner-Mortensen correction applied. Subjects then receive the following drugs, in a randomised fashion, for a period of four weeks each, with BP & ECV measurement at end of each period: doxazosin GITS (Cardura XL) 4 mg b.d.; frusemide 40 mg b.d.; amiloride 5 mg b.d.; placebo.

ELIGIBILITY:
Inclusion Criteria:

* BP >140/85
* 3 antihypertensive drugs (ACE/ARB + calcium channel blocker + thiazide diuretic)

Exclusion Criteria:

* Pregnancy
* Breast Feeding
* Unstable heart failure
* Chronic Liver Disease
* Creatinine >120 mcmol/L
* Contraindication to (or intolerance of) drug used in study
* BP > 180/110

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2003-07; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Change in ECV; change in BP

CONTACTS AND LOCATIONS:
Overall Officials: Timothy WR Doulton, BSc MRCP, Principal Investigator — SGUL
Locations (1):
- Blood Pressure Unit, Dept. Cardiac & Vascular Sciences, SGUL, London, United Kingdom